CLINICAL TRIAL: NCT01721707
Title: Safety and Efficacy to Reduce the IOP of the Fixed Association of Latanoprost 0.005% (50 μg/mL)/ Brinzolamide 1% (10mg/mL) Drops, Compared to Latanoprost 0.005% (50 μg/mL) Drops, in Patients With Open Angle Glaucoma or Ocular Hypertension
Brief Title: Latanoprost/Brinzolamide BID Versus Latanoprost BID in Patients With OAG or OH
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: withdrawn by industry
Sponsor: Adapt Produtos Oftalmológicos Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRINZLAT-12; 08233812.4.0000.5505 (Other: CEP-UNIFESP-PlataformaBrasil)
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: glaucoma; ocular hypertension; latanoprost; brinzolamide
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Latanoprost; brinzolamide; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Latanoprost+Brinzolamide combination (Experimental): Latanoprost 0.005%(50 mg/ml)+brinzolamide 1%(10mg/ml) eye drops
  Interventions: Drug: Latanoprost+Brinzolamide combination
- Latanoprost (Active Comparator): Latanoprost 0.005% (50 mg / ml)
  Interventions: Drug: Latanoprost

INTERVENTIONS:
Drug: Latanoprost+Brinzolamide combination — 1 drop in each eye, 1x/day, at 9PM
  Other Names: Latanoprost 0.005% (50 mg / ml) / brinzolamide 1% (10mg/ml) eye drops
  Arms: Latanoprost+Brinzolamide combination
Drug: Latanoprost — 1 drop in each eye, 1x/day, at 9PM
  Other Names: Latanoprost 0.005% (50 mg / ml)
  Arms: Latanoprost

SUMMARY:
This study is a double-masked, randomized, parallel group study in patients with open angle glaucoma or ocular hypertension.

The aim of this study is to verify the efficacy of the fixed combination of Latanoprost 50 mcg / mL / brinzolamide 10mg/ml eye drops compared to Latanoprost 50μg/mL eye drops in reducing IOP

DETAILED DESCRIPTION:
The study is divided into two sequential phases. The Phase I trial is a Phase Screening / Eligibility, which includes a screening visit, followed by 2 Visits Eligibility (3 visits). The Phase II study is the treatment phase randomized, double-masked that includes visits during therapy at Week 2, Week 6 and Month 3

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older, of either gender and of any race / ethnicity, diagnosed with open angle glaucoma or ocular hypertension, which in the opinion of the investigator does not have enough control with monotherapy or already receiving multiple medications for lowering IOP .
* Patients should be able to understand and sign an informed consent form that has been approved by an Institutional Review Board.
* Measurements of mean IOP in at least 1 eye:

  * ≥ 24 mmHg and ≤ 36 mmHg at timepoint 9am and
  * ≥ 21 mmHg and ≤ 36 mmHg in the 11h timepoint in both Visits Eligibility 1 and after washout of any medication to reduce IOP.
* The mean IOP should not be> 36 mmHg at any timepoint

Exclusion Criteria:

* Fertile women (those not surgically sterile or postmenopausal for at least 1 year) are excluded from study participation if meet any of the following conditions:

  1. currently pregnant or
  2. have tested positive in urine pregnancy Screening Visit or
  3. planning to become pregnant during the study period, or
  4. are breastfeeding, or not using highly effective contraceptive precautions.
* Patients with angle Schaffer Grade <2, as measured by gonioscopy (extreme narrow angle with complete or partial closure).
* Patients with a ratio cup / disc greater than 0.80 (horizontal or vertical).
* Patients presenting with loss of central visual field impairment. The loss of central visual field is defined as a serious sensitivity less than or equal to 10 dB in at least four points of two visual field test closest to the point of attachment.
* Patients who can not safely discontinue use of all medications to ocular IOP reduction for a minimum of 5 days ± 1 day to 28 days ± 1 day prior to Visit E1.
* Chronic inflammatory eye disease, recurrent or severe (ie, scleritis, uveitis, herpetic keratitis).
* Ocular trauma in the past 6 months.
* Eye infection or inflammation of the eye in the last 3 months.
* Retinal disease as clinically significant or progressive retinal degeneration, diabetic retinopathy or retinal detachment.
* Best score corrected visual acuity (BCVA) worse than 55 ETDRS letters (equivalent to approximately 20/80 Snellen).
* Another ocular pathology (including severe dry eye) that may, in the opinion of the investigator, preventing the administration of an alpha-adrenergic agonist and/or an inhibitor of topical carbonic anhydrase (CAI).
* Intraocular surgery within the last 6 months.
* Laser eye surgery in the last 3 months.
* Any abnormality that prevents a reliable applanation tonometry.
* Any other condition including severe illness that would make the patient, in the opinion of the investigator, unsuitable for the study.
* History of cardiovascular disease (eg, coronary heart disease, hypertension, Raynaud's phenomenon, orthostatic hypotension, thromboangiitis), cerebrovascular (eg, cerebral insufficiency), active liver or kidney, severe, unstable or uncontrolled that would prevent the safe administration of an alpha-adrenergic topic or CAI in the opinion of the investigator.

Related to previous or concomitant medications

* Patients with recent use (within 4 weeks of Visit Eligibility 1) salicylate therapy with high dose (> 1 g daily).
* Current or planned treatment with any psychotropic drug that increases the adrenergic response (eg, desipramine, amitriptyline).
* Concomitant use of monoamine oxidase inhibitors.
* Therapy with another investigational agent within 30 days prior to the Screening Visit.
* Hypersensitivity to the drug alpha-adrenergic agonists, oral or topical CAIs, sulfonamide derivatives or any component of the study drugs in the opinion of the investigator.
* Less than 30 days regimen with stable administration before the Screening Visit any medications or substances administered by any route and used chronically that may affect IOP, including among others, β-adrenergic blocking agents.
* Use of ocular hypotensive medication any additional topical or systemic throughout the study.
* Concomitant use of glucocorticoids administered by any route.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
IOP | Month 3
  Change in mean diurnal IOP compared to baseline (Month 3)

SECONDARY OUTCOMES:
IOP changes | week 2, week 6, month 3
  Change in mean IOP from baseline (week 2, week 6, month 3)
IOP measures | week 2, week 6, month 3
  Percentage of patients with IOP <18 mmHg at each visit during therapy and timepoint (week 2, week 6, month 3)

OTHER OUTCOMES:
Biomicroscopy / Fundus examination | Week 2, Week 6, Month 3
  relevant changes observed by physician during biomicroscopy and fundus examination
BCVA | Week 2, Week 6, Month 3
  Decrease of visual acuity observed by BCVA examination

CONTACTS AND LOCATIONS:
Overall Officials: Rubens Belfort Jr, MD, Principal Investigator — Federal University of São Paulo / Hospital São Paulo
Locations (1):
- Department of Ophthalmology / Hospital São Paulo, São Paulo, São Paulo, Brazil